CLINICAL TRIAL: NCT03172052
Title: Evaluating Different Modalities for Pleural Adhesiolysis at Assuit University Hospital
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Montaser Gamal Ahmed, assistent lecturer of Chest Department, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17200064
Record Dates: First submitted 2017-05-21; First posted 2017-06-01 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Pleural Effusion
MeSH Terms: conditions — Pleural Effusion | interventions — Streptokinase; Mesna; Thoracic Surgery, Video-Assisted

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- streptokinase instillation (Experimental): Chemical adhesiolysis by instillation of streptokinase at a dose of 250,000 I.U dissolved in 40 ml of normal saline will be instil in the pleural cavity through the chest tube. we planning to continue the daily instillation as long as the drained fluid volume is >100 cc with a maximum of 14 doses and to stop further instillation if severe complication occurred and if drained fluid through the tube was <100 cc in 24 h provided that tube is patent and properly positioned.
  Interventions: Drug: streptokinase; Drug: MESNA (2-mercaptoethane sulfonate Na); Device: Medical thoracoscopy; Device: Video assisted thoracoscopy (VATS)
- instillation of MESNA (Experimental): Chemical adhesiolysis by instillation of MESNA at a dose of 1800 mg of MESNA i.e. 3 ampoules ( each ampoule contains 3ml and each ml contains 200 mg of MESNA) will be diluted with 20ml of Normal Saline and will be injected into the pleural cavity through the chest tube for three consecutive days.
  Interventions: Drug: streptokinase; Drug: MESNA (2-mercaptoethane sulfonate Na); Device: Medical thoracoscopy; Device: Video assisted thoracoscopy (VATS)
- Medical thoracoscopy procedure (Experimental): Medical thoracoscopy procedure will be carried at endoscopy unit at chest department via, semi rigid thoracoscope
  Interventions: Drug: streptokinase; Drug: MESNA (2-mercaptoethane sulfonate Na); Device: Medical thoracoscopy; Device: Video assisted thoracoscopy (VATS)
- Video assisted thoracoscopy (VATS) (Experimental): Video assisted thoracoscopy (VATS) at cardiothoracic surgery department.
  Interventions: Drug: streptokinase; Drug: MESNA (2-mercaptoethane sulfonate Na); Device: Medical thoracoscopy; Device: Video assisted thoracoscopy (VATS)

INTERVENTIONS:
Drug: streptokinase — • Chemical adhesiolysis by instillation of streptokinase at a dose of 250,000 I.U dissolved in 40 ml of normal saline will be instil in the pleural cavity through the chest tube. we planning to continue the daily instillation as long as the drained fluid volume is >100 cc with a maximum of 14 doses and to stop further instillation if severe complication occurred.
  Other Names: sedonase
Drug: MESNA (2-mercaptoethane sulfonate Na) — • Chemical adhesiolysis by instillation of MESNA at a dose of 1800 mg of MESNA i.e. 3 ampoules ( each ampoule contains 3ml and each ml contains 200 mg of MESNA) will be diluted with 20ml of Normal Saline and will be injected into the pleural cavity through the chest tube for three consecutive days.
Device: Medical thoracoscopy — Medical thoracoscopy procedure will be carried at endoscopy unit at chest department via, semi rigid thoracoscope (LTF; Olympus; Tokyo, Japan).
Device: Video assisted thoracoscopy (VATS) — Video assisted thoracoscopy (VATS) at cardiothoracic surgery department.

SUMMARY:
interventional randomized clinical trial will be done at Assuit University Hospital ( Chest Department and Caridothoracic surgery department ),and all patients presented with complex septate pleural effusion in whom the symptoms excepted to be relieved by pleural fluid drainage will be included in our study within the two next years.

DETAILED DESCRIPTION:
The goal in the management of pleural effusion is to provide symptomatic relief by removing fluid from the pleural space and to allow the treatment of the underlying disease. Despite the improvement in the management options of pleural effusion; intrapleural adhesions remain a significant problem in many patients with pleural disease. The presence of adhesions carry a poor prognostic factor in patients with exudative pleural effusions that it may render the drainage of pleural fluid difficulty inspite of tube being patent and correctly positioned.

Two options are currently available to deal with the problem of pleural adhesions, the first is chemical and the second is mechanical adhesiolysis . Chemical adhesiolysis means lysis of the adhesive bands medically by instillation intrapleural chemical agents e.g. streptokinase, urokinase, tissue plasminogen activator, streptodornase, deoxyribonuclease (human recombinant [hr]DNAase), single-chain urokinase plasminogen activator and the uncommonly used MESNA (2-mercaptoethane sulfonate Na) . Mechanical adhesiolysis means breaking up the adhesive bands and removing it by pulling and dissecting via medical thoracoscope, minimally invasive video assisted thoracoscopy (VATS) or more invasive thoracotomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic pleural effusion in whom the symptoms excepted to be relieved by pleural fluid drainage.
* Presence of intrapleural adhesions as documented sonographically.
* Difficult thoracentesis.
* Failure of satisfactory pleural fluid drainage 24 hours following intercostal tube (ICT) placement provided that the tube was properly positioned and not obstructed.
* Written consent, free and informed.

Exclusion Criteria: patients have contraindications for any of our procedures will be excluded.

* Contraindications for streptokinase instillation i.e. (Previous allergic reaction, bronchopleural fistula, trauma or surgery within 48 hrs, history of hemorrhagic stroke, coagulation defects and previous streptokinase thrombolysis).
* Patients who are unfit for general anaesthesia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-08-01 (Estimated); Primary Completion 2019-06-01 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
measurement of adhesiolysis success | 28 days
  Failure of the procedure: still presence of intra pleural adhesion by chest sonoar.
  Partially successful: incomplete removal of intra pleural adhesions. Successful: complete removal of intra pleural adhesions.